CLINICAL TRIAL: NCT06522854
Title: Oral Sildenafil Citrate to Improve Maternal and Neonatal Outcomes in Low-resource Settings: A Randomized Pilot Feasibility Trial
Brief Title: Oral Sildenafil Citrate to Improve Maternal and Neonatal Outcomes in Low-resource Settings
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Lagos, Nigeria (Other); Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso (Other); Lagos State University (Other); National Health and Medical Research Council, Australia (Other); Mater Medical Research Institute (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Waldemar A. Carlo, Edwin M. Dixon Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UAB-300012809; Dixon Endow Chair/3102800 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Intrapartum Fetal Distress; Neonatal Asphyxia; Intrapartum Asphyxia; Instrumental Delivery; Affecting Fetus
Keywords: Sildenafil citrate
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Double blinded, placebo controlled, 1:1 parallel allocation, randomized feasibility trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator and Outcomes Assessor) The only unmasked person will be the pharmacist who dispenses the study medication--sildenafil 50 mg or identical placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Sildenafil 50mg (Active Comparator): Sildenafil citrate 50mg given orally every eight hours up to 3 doses while mother is in labor
  Interventions: Drug: Sildenafil 50 mg Oral Tablet
- Placebo (Placebo Comparator): Identical-appearing treatment that does not contain the test drug given orally every eight hours up to 3 doses while mother is in labor
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 50 mg Oral Tablet — Sildenafil 50 mg given orally every eight hours up to three times while mother is in labor
  Other Names: Revatio
  Arms: Oral Sildenafil 50mg
Drug: Placebo Oral Tablet — Placebo tablet given orally every eight hours up to three times while mother is in labor
  Arms: Placebo

SUMMARY:
The goal of this feasibility pilot clinical trial is to determine if sildenafil citrate 50mg orally, up to three times during labor, can: 1) reduce perinatal mortality and/or bag and mask ventilation at birth in planned vaginal delivery and 2) reduce the incidence of operative delivery (instrumental vaginal birth or emergency cesarean section) for presumed or suspected fetal distress in up to four facilities of different levels of care in low-resource countries.

The main questions it aims to answer are:

Does sildenafil citrate decrease:

1. the incidence of operative delivery (instrumental vaginal birth or emergency cesarean section) for presumed or suspected fetal distress?
2. the incidence of bag and mask ventilation?
3. the incidence of perinatal mortality?

Researchers will compare sildenafil citrate to a placebo (a look-alike substance that contains no drug) to see if sildenafil works to prevent fetal distress necessitating operative delivery, bag and mask resuscitation at birth, and ultimately, perinatal mortality.

Participants will:

1. Take Sildenafil 50 mg or placebo orally every eight hours during labor (up to 3 doses)
2. Have the (mothers and babies) medical charts reviewed for outcomes, including fetal distress, operative delivery, maternal side effects, neonatal bag & mask ventilation, Apgar Scores, and seizures.
3. Have a neonatal neurological assessment prior to discharge
4. Receive telephone call assessments for re-hospitalization or mortality 7 days post delivery

The results of this feasibility pilot trial will be used to inform the design and conduct of a large pragmatic randomized controlled trial to determine if sildenafil citrate, compared to placebo, will decrease fetal distress and perinatal asphyxia.

DETAILED DESCRIPTION:
Pregnant women with planned vaginal deliveries will be screened for eligibility. After informed consent obtained, subjects will be randomly assigned (using computer generated, stratified randomization codes by the pharmacy) to either the treatment arm (Sildenafil citrate) or the placebo concurrent control. Clinicians, researchers, and primary caregivers will be masked. Eligible women will be randomized to receive sildenafil 50 mg orally every 8 hours up to a total of 3 doses or to receive the placebo every 8 hours up to a total of 3 does during the course of labor. Neither medication no placebo will be given following completion of labor. All additional care of the mother and infant will be provided according to the local standard of care. A neurological examination (Sarnat and Thompson) will be completed on the infant within 24 hours after birth. Neonatal oxygen saturation will be measured by pulse oximetry at 48 hours or discharge, whichever comes first. Outcomes will be collected following delivery, discharge, and 7-days post-partum. 7-day follow-up for outcomes will be obtained via a telephone call.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women presenting in early labor with a term pregnancy (≥ 37 weeks to 41wks 6days gestation )

   * Early labor will be defined as cervical dilation less than 7cm
   * Gestational age will be calculated from the most reliable variable using the following hierarchy of reliability: 2) gestational dating ultrasound completed at any time during the pregnancy (with preference to the earliest exam); 2) date of last menstrual period if menses are regular.
2. Planned vaginal delivery and admission to health facility with clear plan for spontaneous or induced vaginal delivery
3. Maternal age ≥ 18yrs

Exclusion Criteria:

1. Unknown gestational age
2. Non-cephalic fetal presentation
3. Plan for cesarean delivery prior to enrollment
4. Previous uterine scar (cesarean section and/or myomectomy)
5. Advanced stage of labor (7 cm or greater cervical dilation per local standards) and pushing, or too distressed to understand, confirm, or give informed consent regardless of cervical dilation
6. Not capable of giving consent due to other health problems, such as obstetric emergencies (i.e. antepartum hemorrhage) or mental disorder
7. Maternal contraindication to sildenafil therapy, such as hypersensitivity to nitrates or nitrites
8. Recognized major structural fetal anomaly
9. Previous randomization in the trial

Ages: 0 Days to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of perinatal mortality | 96 hours after enrollment
  Documentation of stillbirth or neonatal death
Percentage of use of bag and mask in neonates after delivery | 20 minutes after delivery
  Documentation of the use of bag and mask ventilation as resuscitation after delivery
Percentage of operative delivery | 96 hours after enrollment
  Documentation of type of delivery
Indication for operative delivery | 96 hours after enrollment
  Documentation of type of delivery

SECONDARY OUTCOMES:
Percentage of mothers who received fetal heart rate monitoring | 96 hours after enrollment
  Documentation of rate of heart rate monitoring
Indication for fetal heart rate monitoring | 96 hours after enrollment
  Documentation of the indication for use of fetal heart rate monitoring
Apgar Score | 1 minute and 5 minutes after birth
  Documentation of Apgar score at 1 minute and 5 minutes (Value 0-10, with 10 meaning better outcome)
Percentage of neonates with neonatal encephalopathy by Sarnat Score | 24 hours after birth
  Documentation of neonatal neurological exam determined by "modified Sarnat Score (no, mild, moderate, and severe"; higher score indicates more encephalopathy
Percentage of neonates with neonatal encephalopathy by Thompson Score | 24 hours after birth
  Documentation of neonatal neurological exam determined by "Thompson Score (no, mild, moderate, and severe)"; higher score indicates more severe encephalopathy
Percentage of infants with neonatal hypoxic-ischemic encephalopathy | 96 hours after enrollment
  Documentation of neonatal encephalopathy
Percentage of neonates with hypoxemia | 48 hours after birth or at discharge, if early discharge
  Documentation of saturations < 95% measured by noninvasive pre/post pulse oximetry
Percentage of neonatal ICU admissions | 96 hours after enrollment
  Documentation of admission to the Neonatal Intensive Care Unit or comparable level of care
Percentage of maternal rehospitalization | 7 days
  Maternal rehospitalization after initial discharge from the hospital assessed by telephone call to mother
Percentage of neonatal rehospitalization | 7 days
  Neonatal rehospitalization after initial discharge from the hospital assessed by telephone call to mother

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- Nigeria (4):
  - Lagos Island Maternity Hospital, Lagos, Lagos
  - University Teaching Hospital, University of Lagos, Lagos, Lagos
  - Mother and Child Hospital, Surulere, Lagos
  - Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso, Oyo State